CLINICAL TRIAL: NCT01083303
Title: A Randomized Trial of Weaning Preterm Infants at 1500g From Incubators: Effect on Failure to Wean, Weight Gain and Energy Expenditure
Brief Title: Weaning Preterm Infants at 1500 Grams From Incubators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TASMC08BI05089CTIL
Record Dates: First submitted 2009-07-02; First posted 2010-03-09 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Preterm Infants
Keywords: energy expenditure; hypothermia; body temperature; weaning; preterm infants
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- weaning at 1500 g (Experimental): weaning infants from an incubator at 1500 g
  Interventions: Behavioral: Weaning Preterm Infants from an incubator
- weaning at 1600 g (Active Comparator): weaning infants from an incubator at 1600 g
  Interventions: Behavioral: Weaning Preterm Infants from an incubator

INTERVENTIONS:
Behavioral: Weaning Preterm Infants from an incubator — Eligible infants are to be randomized by computer generated random numbers to either the study group weaned at 1500 gr. or the control group weaned at 1600 gr. Both groups were weaned to a warming bassinet.

SUMMARY:
Background: The weight at which infants are weaned from incubators varies among neonatal units.

Objective: To determine the effect on weight gain, temperature stability and resting energy expenditure (REE) of weaning infants at body weight of 1500 g versus 1600 g.

Design/Methods: infants will be randomized to incubator weaning at the weight of 1500 g or 1600 g. Preterm infants 1500 g birth weight, fully enterally fed, and without supplemental oxygen, at the postnatal age of 2 weeks will be included. Infants will be weaned to a warming bassinet (Babytherm 8000, Dräger) set to keep a mattress temperature of 37°C while decreasing it gradually to room temperature. Failure to wean is defined as core body temperature of < 36.1°C. Data collection included skin and rectal temperature obtained before weaning, and at 1/2, 1, 2, 6, 24, and 48 hours after weaning, weekly weight gain (g/kg/d). REE (kcal/kg/24h) will be measured by indirect calorimetry (Deltatrac II, Finland) before and 24 hours after weaning.

DETAILED DESCRIPTION:
Eligible infants will be randomized by computer generated random numbers, to either the study group weaned at 1500 g or the control group weaned at 1600 g. Both groups will be weaned to a warming bassinet (Babytherm 8000, Drager). The Babytherm 8000 WB is an open care infant warming system with a warmed gel mattress with temperature control . The system is set to keep the mattress temperature of 37 degrees Celsius while decreasing it gradually to 32 0C and shutting the system off. On transfer to the Babytherm infants are dressed with a hat and two vests. Only after the infant maintained a normal body temperature under these conditions he could be transferred to an open bassinet. Failure to wean was defined as core body temperature of <36.10C.

Data collection included skin and rectal temperature obtained before weaning, and at 1/2, 1, 2, 6, 24, and 48 hours after weaning, daily and weekly weight gain (g/kg/d). Resting Energy Expenditure- REE (kcal/kg/24h) is measured by indirect calorimetry (Deltatrac II, Finland) before and 24 hours after weaning to the warming bassinet.

Data Collection included: PR temperature after 30 min, 60 min, 2 hours, 6 hours, 24 hours, after which temperatures were taken 4-hourly until 48 hours (degrees C), skin (axillary) temperature (degrees C), after 30 min, 60 min, 2 hours, 6 hours, and than again every 4 hours until 48 hours. REE (kcal/kg/24h)rate of hypothermia requiring return to the incubator, weight gain after 24 hours of weaning and over 1 week.( g/kg/d),time to discharge ( days).

ELIGIBILITY:
Inclusion Criteria:

* stable preterm infants weighing ≤1500 g
* fully enterally fed, and without supplemental oxygen
* steroid or antibiotics treatment
* at the postnatal age of ≥ 2 weeks were included
* infants < than 2 weeks of age

Exclusion Criteria:

* ventilated infants or those requiring oxygen supplementation
* parenteral nutrition
* antibiotic treatment or steroids treatment were excluded

Min Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
successful and safe weaning from convective incubator of stable preterm infants to a warming bassinet at body weight of 1500g compared with 1600g. | Ten days

SECONDARY OUTCOMES:
Resting energy expenditure REE (kcal/kg/24h) measurements | Fourty eight hours

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Dollberg, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Neonatology department Tel Aviv Medical Center, Tel Aviv, Israel